CLINICAL TRIAL: NCT05705830
Title: A Multicenter Randomized Controlled Study of Pulse Magnetotherapy Combined Medication in the Treatment of Patients With Anxiety Disorder and Insomnia
Brief Title: A Multicenter Randomized Controlled Study of Pulse Magnetotherapy Combined Medication in Anxiety Combined With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0704
Record Dates: First submitted 2022-10-25; First posted 2023-01-31 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-10

CONDITIONS: Anxiety Disorder; Insomnia
Keywords: Anxiety; Insomnia; Pulse Magnetotherapy
MeSH Terms: conditions — Anxiety Disorders; Sleep Initiation and Maintenance Disorders | interventions — Selective Serotonin Reuptake Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pulse Magnetotherapy+medication group (Experimental): 150 patients with anxiety disorder and insomnia who met the inclusion criteria received pulse magnetic therapy and conventional antianxiety drugs
  Interventions: Device: Pulse magnetic therapy; Drug: Selective serotonin reuptake inhibitors （SSRI）
- medication group (Sham Comparator): 150 patients with anxiety disorder and insomnia who met the inclusion criteria received sham magnetic therapy and conventional antianxiety drugs
  Interventions: Drug: Selective serotonin reuptake inhibitors （SSRI）; Device: Shame magnetic therapy
- Healthy control (Other): 100 healthy controls who met the inclusion criteria received sham magnetic therapy
  Interventions: Device: Shame magnetic therapy

INTERVENTIONS:
Device: Pulse magnetic therapy — Pulse magnetic therapy SM-II (2019102133903)
  Arms: Pulse Magnetotherapy+medication group
Drug: Selective serotonin reuptake inhibitors （SSRI） — Anti-anxiety Drugs
  Arms: Pulse Magnetotherapy+medication group; medication group
Device: Shame magnetic therapy — Shame magnetic therapy
  Arms: Healthy control; medication group

SUMMARY:
The goal of this clinical trial is to explore the therapeutic effect of pulse magnetic therapy system combined with drug therapy on patients with anxiety and insomnia. The main questions it aims to answer are:

1. Whether the pulse magnetic therapy system is benefit on improving insomnia in anxiety patients.
2. This improvement is not due to the placement of the instrument。 Participants will accept pulse magnetic therapy (stimulation/sham stimulation) and accept scale evaluation before and after treatment.

Researchers will compare the pulse magnetic stimulation group, sham stimulation group and healthy controls to see if the pulse magnetic stimulation do effect on insomnia of anxiety patients.

DETAILED DESCRIPTION:
Insomnia is the most common symptom of anxiety disorder, which has an important impact on the prognosis of anxiety. Pulse magnetic therapy system, with its advantages of compact, convenient, easy to carry, and not limited by the scene and time, has gradually become a common tool for sleep monitoring and treatment. This study is a multicenter randomized controlled design, including 150 cases in the pulse magnetic stimulation+drug treatment group, 150 cases in the sham pulse magnetic stimulation+drug treatment group and 100 healthy controls. Before and after treatment, the patients were comprehensively measured and evaluated with Insomnia Severity Index (ISI), Hamilton Depression Rating Scale 17 (HAMD), Hamilton Anxiety Rating Scale (HAMA), Pittsburgh Sleep Quality Index (PSQI), Self-Rating Sleep Scale (SSRS), Self-Rating Symptom Scale 90 (SCL-90), Quality of Life Scale (SF-36), and Treatment Adverse Reaction Scale (TESS), and sleep monitoring was conducted at the same time, To explore the therapeutic effect of pulse magnetic therapy system detector combined with drug therapy on patients with anxiety and insomnia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who met the diagnostic criteria for anxiety disorder in the Diagnostic and Statistical Manual of Mental Disorders (Fifth edition; DSM-5) and were accompanied by insomnia with 14 <HAMA<21 , HAMD<17 , and PSQI>7 ;
2. Education level is unlimited;
3. Age: 18-55 years old.

Exclusion Criteria:

1. Have bipolar disorder, schizophrenia, depression and other mental diseases;
2. Have a clear history of head trauma, alcoholism, brain tumors, diabetes, hypertension, and serious primary heart, liver, kidney, and blood system diseases;
3. At present, patients with sleep disorders are being treated by other means besides drugs;
4. Pregnant and lactating women;
5. Have a history of seizures or strong positive family history of epilepsy;
6. Implantation of cardiac pacemaker;
7. Those receiving deep brain stimulation treatment;
8. There are metal or magnetic implants in the body (including but not limited to the brain);
9. Participated in clinical trials of other drugs and medical devices in recent 3 months;
10. Other researchers believe that they do not meet the conditions for inclusion.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Change value of insomnia severity index (ISI) from baseline in the fourth week of intervention
  Insomnia Severity Index total score reduction>50%, the range of Insomnia Severity Index total score is 0-28.

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Lin, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - Changxing County People's Hospita, Changxing, Zhejiang
  - Linping First People's Hospital, Linping, Zhejiang
  - The Fourth Affiliated Hospital of Zhejiang University School of medicine, Yiwu, Zhejiang